CLINICAL TRIAL: NCT06206616
Title: Liver Steatosis in Pediatric Celiac Disease Patients: Exploring the Epidemiological and Pathophysiological Features of an Underestimated Condition
Brief Title: Liver Steatosis in Pediatric CD Patients
Status: Not yet recruiting | Type: Observational
Sponsor: University of Palermo (Other)
Collaborators: ARNAS Civico Di Cristina Benfratelli Hospital (Other); Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello (Other)
Responsible Party: Principal Investigator, Aurelio Seidita, Assistant Professor, University of Palermo
Other Study IDs: ASAC01
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-12

CONDITIONS: Celiac Disease in Children; Non-Alcoholic Fatty Liver Disease
Keywords: Celiac Disease; Non-Alcoholic Fatty Liver Disease; Intestinal Permeability; Inflammatory Cytokines; Children
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Celiac Disease | interventions — Diet, Gluten-Free

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Celiac Disease Children: Pediatric patients affected by newly diagnosed CD according to the European Society for Paediatric Gastroenterology Hepatology and Nutrition (ESPGHAN) criteria will be evaluated before the start of gluten-free diet and after 6 months of gluten-free diet.
  Interventions: Behavioral: Gluten-free diet

INTERVENTIONS:
Behavioral: Gluten-free diet — Pediatric patients affected by newly diagnosed Celiac Disease (CD) according to the European Society for Paediatric Gastroenterology Hepatology and Nutrition (ESPGHAN) criteria will start a gluten-free diet (GFD), as normally expected for all CD patients. The assessment of adherence to the GFD will be carried out through the monthly compilation, by the children and/or their parents, of a specifically created and validated questionnaire.
  Before and after the start of GFD enrolled patients will undergo an abdominal ultrasound to establish the presence and degree of hepatic steatosis.

SUMMARY:
Celiac disease (CD) is an autoimmune enteropathy triggered by the intake of gluten, characterized by a genetic predisposition. Although, CD is often associated with malabsorption symptoms, a growing number of affected subjects are overweight or frankly obese. One of the conditions that is most frequently detected in pauci/asymptomatic subjects is an increase in transaminases, which often regresses completely after the start of GFD.

More recently, a specific liver disorder has shown a certain relevance in adult patients suffering from CD, so much so that the European Society for the Study of Coeliac Disease (ESsCD) has cited it among the possible comorbidities which should be screened in CD subjects: Non-Alcoholic Fatty Liver Disease (NAFLD).

In adults, a non-random association between CD and NAFLD has been demonstrated, showing a CD prevalence rate of 2-14% among patients with NAFLD. Few studies have focused on this same aspect in pediatric age, reporting contrasting data.

Several factors have been advocated as putative responsible of association between CD and NAFLD: dietary imbalances, intestinal mucosa permeability impairment, alterations of the intestinal microbiota.

The objectives of this study are:

1. define, retrospectively, the prevalence of NAFLD in a pediatric population affected by CD and study its possible association with GFD.
2. define the possible role of the intestinal permeability alteration and/or the intestinal mucosa damage and/or the proinflammatory status in the development of NAFLD in children affected by CD.

DETAILED DESCRIPTION:
Background Celiac disease (CD), an autoimmune enteropathy triggered by the intake of gluten, is a widespread pathology, with a worldwide estimated prevalence of approximately 1%, characterized by both gastrointestinal and systemic symptoms, both in adults and children, which are usually resolved by eliminating gluten from the diet (Gluten-Free Diet, GFD). However, it still remains an under-diagnosed condition (to date the overall prevalence in Italy is 0.37% and in Sicily 0.35%).

Although, CD is often associated with malabsorption symptoms (steatorrhea, weight loss, nutritional deficits, etc.), a growing number of affected subjects are overweight or frankly obese. One of the conditions that is most frequently detected in pauci/asymptomatic subjects is an increase in transaminases, which often regresses completely after the start of GFD.

More recently, a specific liver disorder has shown a certain relevance in patients suffering from CD, so much so that the European Society for the Study of Coeliac Disease (ESsCD) has cited it among the possible comorbidities which should be screened in CD subjects: Non-Alcoholic Fatty Liver Disease (NAFLD). This condition affects approximately 34% of overweight or frankly obese children and is closely related, both in children and adults, to the traits of metabolic syndrome, so much so that today it is preferably referred to as Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD). In adults, a non-random association between CD and NAFLD has been demonstrated, showing a CD prevalence of 2-14% among patients with NAFLD. Few studies have focused on this same aspect in pediatric age, however reporting that the prevalence of CD among children with NAFLD could be comparable to the prevalence of CD in the general pediatric population. Nevertheless, a study conducted on 11488 children (0-19 years) affected by CD compared with 57029 healthy children supports the hypothesis of a close association between CD and NAFLD in childhood. Authors proved a 4.6 relative risk value of NAFLD in CD patients.

Several factors have been advocated as putative responsible for this association: 1) dietary imbalances due to the adoption of GFD, rich in fats and sugars and low in fiber; 2) alteration of intestinal permeability, with an increase in the translocation of bacterial substances from the gut, which, are transported directly to the liver, where they are able to generate inflammatory processes mediated by the nuclear factor kappa-light-chain-enhancer of activated B cells (NF-kB), activated by the Tool-like receptor 4 (TLR4)-Lipopolysaccharide (LPS)-LPS Binding Protein (LPB) complex, with production of proinflammatory cytokines [Tumor Necrosis Factor (TNF)-α, Interleukine (IL)-1β, IL-6, IL-12, IL-18); 3) alterations of the intestinal microbiota.

Objectives

Primary objective: define, retrospectively, the prevalence of NAFLD in a pediatric population affected by CD and study its possible association with GFD:

Objective 1.1: identify the prevalence of NAFLD before the introduction of the GFD in an already diagnosed pediatric celiac; Objective 1.2: identify the prevalence of NAFLD after at least 12 months of GFD in an already diagnosed pediatric celiac; Objective 1.3: compare the prevalence of NAFLD before and after (at least 12 months) the introduction of the GFD in all pediatric celiac patients for whom both pre- and post-GFD data are available; Objective 1.4: establish a possible correlation between the presence/absence of NAFLD, both before and after the adoption of the GFD, and clinical, laboratory, immunological, genetic and histological parameters, in order to identify a subgroup of celiac children potentially predisposed to the NAFLD development; Objective 1.5: establish any changes in the clinical, laboratory, immunological, genetic and histological parameters of the population referred to in objective 1.3 and establish whether there is a correlation between these and the possible onset/regression of NAFLD.

Secondary objective: define the possible role of the intestinal permeability alteration and/or the intestinal mucosa damage and/or the proinflammatory status in the development of NAFLD in children affected by CD:

Objective 2.1: identify the possible presence of serological markers of altered intestinal permeability and/or intestinal mucosa damage in a population of celiac children prospectively enrolled at the Pediatric Clinic of the Children's Hospital "G. Di Cristina" before the start of the GFD (T0).

Objective 2.2: Identify the possible presence of blood markers of inflammation in the population referred to in point 2.1 at T0.

Objective 2.3: define the existence of an association between the markers of altered intestinal permeability and/or mucosal damage and/or inflammation and the presence of NAFLD in the population referred to in point 2.1 at T0.

Objective 2.4: evaluate any changes in serological markers of altered intestinal permeability and/or mucosal damage in the population referred to in point 2.1 after 6 months of strict adherence to the GFD (T1).

Objective 2.5: evaluate any changes in blood markers of inflammation in the population referred to in point 2.1 at T1.

Objective 2.6: define the existence of an association between the markers of altered intestinal permeability and/or mucosal damage and/or inflammation and the presence of NAFLD in the population referred to in point 2.1 at T1.

Materials and methods Primary objective To achieve the primary objective of the study, all the medical records of pediatric patients suffering from CD already diagnosed according to the European Society for Paediatric Gastroenterology Hepatology and Nutrition (ESPGHAN) criteria at the Pediatric Clinic of the Children's Hospital "G. Di Cristina" will be retrospectively analyzed.

Objectives 1.1, 1.2 and 1.3 To achieve objectives 1.1 and 1.2, the presence and degree of steatosis diagnosed by abdominal ultrasound will be assessed before the start of the GFD (objective 1.1) or after at least 12 months from the introduction of the GFD (objective 1.2).

To achieve objective 1.3, a sub-analysis of the presence and degree of steatosis will be performed in all those patients who have undergone an abdominal ultrasound both before and after the introduction of GFD.

Objectives 1.4 and 1.5 To achieve objective 1.4, clinical (sex, ethnicity, age at diagnosis, BMI, symptoms, duration of GFD), laboratory (transaminasemia, albuminemia, total cholesterolemia and subclasses, triglyceridemia, fasting glycemia, insulinemia, Homeostasis Model Assessment-Insulin Resistance HOMA-IR Index), immunological [anti-gliadin antibodies (AGA), anti-tissue transglutaminase antibodies (tTG), anti-endomysial antibodies (EMA)], genetic (HLA structure) and histological (Marsh duodenal histological classification, presence of eosinophilic infiltration, etc.) data of all included patients will be collect, both before (target population 1.1) and after (target population 1.2) the introduction of the GFD.

To achieve objective 1.5, the same clinical, laboratory, immunological, genetic and histological parameters analyzed for objective 1.4 will be analyzed, if available both before and after the introduction of the GFD, in order to establish whether there is a correlation between these and the possible onset/regression of NAFLD in the population referred to in objective 1.3.

Secondary objective To achieve the secondary objective of the study, pediatric patients affected by newly diagnosed CD according to the ESPGHAN criteria will be prospectively enrolled at the at the Pediatric Clinic of the Children's Hospital "G. Di Cristina". The number of subjects to be enrolled will be equal to 91, considering, in the Province of Palermo, Sicily, Italy, a pediatric population (between 0 and 14 years) of 170,468 subjects, a prevalence of CD equal to 1%, a confidence level of 95% and a confidence interval of 10%. Furthermore, as the exact prevalence of NAFLD in children with CD it's not clearly defined, results derived from the retrospective part of this study (objective 1.1) will be used to maintain a proportion between subjects enrolled without and with pre-GFD NAFLD ("competitive enrollment").

Objectives 2.1, 2.2, 2.3 To achieve objective 2.1, all enrolled subjects, for whom the same clinical, laboratory, immunological, genetic and histological parameters analyzed for objective 1.4 must be available (the latter only if necessary for diagnosis), in order to make a comparison possible, will be subjected to blood sampling for the identification of serological markers of altered intestinal permeability [zonulin (Zo), occludin (OCLN), anti-OCLN antibodies, claudin 1 (CLDN1) and anti-CLDN1 antibodies] and mucosal damage [Intestinal Fatty Acid Binding Protein 2 (iFABP2)], lipopolysaccharide (LPS), lipopolysaccharide binding protein (LPB)] before starting the GFD (T0). The blood sampling will coincide with the one necessary for the diagnostic definition of the patient's clinical picture.

To achieve objective 2.2, all enrolled subjects will undergo a blood sample before starting the GFD (T0), for the identification of the following inflammatory markers: TNF-α, IL-1β, IL-6, IL-12, IL-18. The blood sampling will coincide with the one necessary for the diagnostic definition of the patient's clinical picture.

To achieve objective 2.3, all enrolled subjects, before starting the GFD (T0), will undergo an abdominal ultrasound to study hepatic steatosis according to the methods previously described and a statistical correlation analysis will be carried out between the presence/absence of NAFLD and the markers assayed for objective 2.1 and 2.2.

The assay of intestinal permeability and mucosal damage markers will be carried out using the ELISA method, with commercially available kits, following the manufacturers' instructions.

The measurement of inflammation markers will be performed by intracellular staining with flow cytometric method on peripheral blood mononuclear cells (PBMC) extracted from patients' blood samples.

Objectives 2.4, 2.5, 2.6 To achieve objective 2.4, all enrolled subjects, for whom the same clinical, laboratory and immunological parameters analyzed at T0 must be available, in order to make a comparison possible, will be subjected to a blood sample for the identification of serological markers of altered intestinal permeability and mucosal damage already measured at T0 (see objective 2.1), after 6 months of strict adherence to the GFD (T1). The blood sampling will coincide with the one necessary to re-evaluate the patient's clinical picture after 6 months of adherence to the GFD.

To achieve objective 2.5, all enrolled subjects will undergo a blood sample to identify the inflammation markers already dosed at T0 (see objective 2.2), after 6 months of strict adherence to the GFD (T1). The blood sampling will coincide with the one necessary to re-evaluate the patient's clinical picture after 6 months of adherence to the GFD.

To achieve objective 2.6, all enrolled subjects, after 6 months of strict adherence to the GFD (T1), will undergo abdominal ultrasound to study hepatic steatosis according to the methods previously described and a statistical correlation analysis will be carried out between the presence/absence of NAFLD and the markers assayed for objective 2.4 and 2.5.

The assessment of adherence to the GFD will be carried out through the monthly compilation, by the children and/or their parents, of a specifically created and validated questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age >1 and <14 years
* Celiac Disease diagnosis according European Society for Paediatric Gastroenterology Hepatology and Nutrition (ESPGHAN) criteria

Exclusion Criteria:

* age <1 and >14 years;
* self-exclusion of gluten/wheat from the diet and refusal to reintroduce it, for diagnostic purposes, before entering the study;
* bacterial and/or parasitic infections;
* diagnosis of chronic inflammatory intestinal diseases and other organic pathologies affecting the digestive system (for example, serious liver diseases), nervous system diseases, immunological deficits and impairments that limit physical activity;
* diagnosis of cancer
* patients undergoing chemotherapy and/or radiotherapy.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Celiac Disease diagnosis according European Society for Paediatric Gastroenterology Hepatology and Nutrition (ESPGHAN) criteria, aged 1-14 years.
Sampling Method: Probability Sample
Enrollment: 91 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Historical Nonalcoholic Fatty Liver Disease Prevalence in Pediatric Celiac Disease Patients before Gluten Free Diet | Retrospective (years 2000-2023)
  We will review all the clinical charts of historical Celiac Disease pediatric patients to identify the number of patients suffering from Nonalcoholic Fatty Liver Disease before the start of gluten free diet.
  Hepatic steatosis will be ascertained by ultrasound examination and classified as follows: absent (score 0), present (score 1)
Historical Nonalcoholic Fatty Liver Disease Prevalence in Pediatric Celiac Disease Patients after Gluten Free Diet | Retrospective (years 2000-2023)
  We will review all the clinical charts of historical Celiac Disease pediatric patients to identify the number of patients suffering from Nonalcoholic Fatty Liver Disease after the start of gluten free diet (at least 1 year of diet).
  Hepatic steatosis will be ascertained by ultrasound examination and classified as follows: absent (score 0), present (score 1)
Historical Nonalcoholic Fatty Liver Disease Degree in Pediatric Celiac Disease Patients before Gluten Free Diet | Retrospective (years 2000-2023)
  We will review all the clinical charts of historical Celiac Disease pediatric patients to identify the steatosis degree of patients suffering from Nonalcoholic Fatty Liver Disease before the start of gluten free diet.
  Hepatic steatosis will be ascertained by ultrasound examination and classified as follows: when the echostructure of the liver is normal; mild (score 1 = mild), when there is a mild and diffuse increase in hepatic echogenicity, with normal visualization of the portal vein wall and diaphragm; moderate (score 2 = moderate), in case of moderate increase in hepatic echogenicity, with slightly altered appearance of the portal vein wall and diaphragm; severe (score 3 = severe), in case of marked increase in hepatic echogenicity, with poor or absent visualization of the wall of the portal vein, the diaphragm and the posterior part of the right hepatic lobe
Historical Nonalcoholic Fatty Liver Disease Degree in Pediatric Celiac Disease Patients after Gluten Free Diet | Retrospective (years 2000-2023)
  We will review all the clinical charts of historical Celiac Disease pediatric patients to identify the steatosis degree of patients suffering from Nonalcoholic Fatty Liver Disease after the start of gluten free diet (at least 1 year of diet).
  Hepatic steatosis will be ascertained by ultrasound examination and classified as follows: when the echostructure of the liver is normal; mild (score 1 = mild), when there is a mild and diffuse increase in hepatic echogenicity, with normal visualization of the portal vein wall and diaphragm; moderate (score 2 = moderate), in case of moderate increase in hepatic echogenicity, with slightly altered appearance of the portal vein wall and diaphragm; severe (score 3 = severe), in case of marked increase in hepatic echogenicity, with poor or absent visualization of the wall of the portal vein, the diaphragm and the posterior part of the right hepatic lobe
Historical Nonalcoholic Fatty Liver Disease Prevalence Change in Pediatric Celiac Disease Patients | Retrospective (years 2000-2023); 1 year of diet
  A comparison between pre and post gluten free diet (1 year of diet) Nonalcoholic Fatty Liver Disease evidence will be performed in all historical pediatric celiac disease patients who have undergone an abdominal ultrasound both before and after the introduction of the GFD. Hepatic steatosis will be ascertained by ultrasound examination and classified as follows: absent (score 0), present (score 1).
  Difference will be considered significant for p<0.05.
Historical Nonalcoholic Fatty Liver Disease Degree Change in Pediatric Celiac Disease Patients | Retrospective (years 2000-2023); 1 year of diet
  A comparison between pre and post gluten free diet (1 year of diet) Nonalcoholic Fatty Liver Disease degree will be performed in all historical pediatric celiac disease patients who have undergone an abdominal ultrasound both before and after the introduction of the GFD.
  Hepatic steatosis will be ascertained by ultrasound examination and classified as reported in outcomes 3 and 4.
  Difference will be considered significant for p<0.05.

SECONDARY OUTCOMES:
Historical Aspartate Aminotransferase changes between pre and post gluten free diet in Nonalcoholic Fatty Liver Disease Pediatric Celiac Disease Patients | Retrospective (years 2000-2023); 1 year of diet
  Aspartate Aminotransferase will be assessed in all historical subjects who had or did not have a change in liver steatosis degree between pre and post 1 year of gluten free diet.
  Difference will be considered significant for p<0.05.
Historical Alanine Aminotransferase changes between pre and post gluten free diet in Nonalcoholic Fatty Liver Disease Pediatric Celiac Disease Patients | Retrospective (years 2000-2023); 1 year of diet
  Alanine Aminotransferase will be assessed in all historical subjects who had or did not have a change in liver steatosis degree between pre and post 1 year of gluten free diet. Difference will be considered significant for p<0.05.
Historical Albuminemia changes between pre and post gluten free diet in Nonalcoholic Fatty Liver Disease Pediatric Celiac Disease Patients | Retrospective (years 2000-2023); 1 year of diet
  Albuminemia will be assessed in all historical subjects who had or did not have a change in liver steatosis degree between pre and post 1 year of gluten free diet. Difference will be considered significant for p<0.05.
Historical total cholesterolemia changes between pre and post gluten free diet in Nonalcoholic Fatty Liver Disease Pediatric Celiac Disease Patients | Retrospective (years 2000-2023); 1 year of diet
  Total cholesterolemia will be assessed in all historical subjects who had or did not have a change in liver steatosis degree between pre and post 1 year of gluten free diet. Difference will be considered significant for p<0.05.
Historical fasting glycemia changes between pre and post gluten free diet in Nonalcoholic Fatty Liver Disease Pediatric Celiac Disease Patients | Retrospective (years 2000-2023); 1 year of diet
  Fasting glycemia will be assessed in all historical subjects who had or did not have a change in liver steatosis degree between pre and post 1 year of gluten free diet. Difference will be considered significant for p<0.05.
Historical insulinemia changes between pre and post gluten free diet in Nonalcoholic Fatty Liver Disease Pediatric Celiac Disease Patients | Retrospective (years 2000-2023); 1 year of diet
  Insulinemia will be assessed in all subjects who had or did not have a change in liver steatosis degree between pre and post 1 year of gluten free diet. Difference will be considered significant for p<0.05.
Historical Homeostasis Model Assessment-Insulin Resistance (HOMA-IR) changes between pre and post gluten free diet in Nonalcoholic Fatty Liver Disease Pediatric Celiac Disease Patients | Retrospective (years 2000-2023); 1 year of diet
  HOMA-IR Index will be assessed in all historical subjects who had or did not have a change in liver steatosis degree between pre and post 1 year of gluten free diet. Difference will be considered significant for p<0.05.
Historical anti-gliadin immunoglobulin A changes between pre and post gluten free diet in Nonalcoholic Fatty Liver Disease Pediatric Celiac Disease Patients | Retrospective (years 2000-2023); 1 year of diet
  Anti-gliadin immunoglobulin A will be assessed in all historical subjects who had or did not have a change in liver steatosis degree between pre and post 1 year of gluten free diet. Difference will be considered significant for p<0.05.
Historical anti-gliadin immunoglobulin G changes between pre and post gluten free diet in Nonalcoholic Fatty Liver Disease Pediatric Celiac Disease Patients | Retrospective (years 2000-2023); 1 year of diet
  Anti-gliadin immunoglobulin G will be assessed in all historical subjects who had or did not have a change in liver steatosis degree between pre and post 1 year of gluten free diet. Difference will be considered significant for p<0.05.
Historical anti-tissue transglutaminase immunoglobulin A changes between pre and post gluten free diet in Nonalcoholic Fatty Liver Disease Pediatric Celiac Disease Patients | Retrospective (years 2000-2023); 1 year of diet
  Anti-tissue transglutaminase immunoglobulin A will be assessed in all historical subjects who had or did not have a change in liver steatosis degree between pre and post 1 year of gluten free diet. Difference will be considered significant for p<0.05.
Historical anti-tissue transglutaminase immunoglobulin G changes between pre and post gluten free diet in Nonalcoholic Fatty Liver Disease Pediatric Celiac Disease Patients | Retrospective (years 2000-2023); 1 year of diet
  Anti-tissue transglutaminase immunoglobulin G will be assessed in all historical subjects who had or did not have a change in liver steatosis degree between pre and post 1 year of gluten free diet. Difference will be considered significant for p<0.05.
Historical anti-endomysial antibodies immunoglobulin A changes between pre and post gluten free diet in Nonalcoholic Fatty Liver Disease Pediatric Celiac Disease Patients | Retrospective (years 2000-2023); 1 year of diet
  Anti-endomysial antibodies immunoglobulin A will be assessed in all historical subjects who had or did not have a change in liver steatosis degree between pre and post 1 year of gluten free diet. Difference will be considered significant for p<0.05.
Historical human leukocyte antigen status in Nonalcoholic Fatty Liver Disease Pediatric Celiac Disease Patients | Retrospective (years 2000-2023)
  Human leukocyte antigen status will be assessed in all subjects who had or did not have a change in liver steatosis degree between pre and post 1 year of gluten free diet. Difference will be considered significant for p<0.05.
Historical Marsh duodenal histological classification changes between pre and post gluten free diet in Nonalcoholic Fatty Liver Disease Pediatric Celiac Disease Patients | Retrospective (years 2000-2023); 1 year of diet
  Marsh duodenal histological classification will be assessed in all historical subjects who had or did not have a change in liver steatosis degree between pre and post 1 year of gluten free diet, and who underwent gastroscopy both before and after start of gluten-free diet. Difference will be considered significant for p<0.05.
Duodenal eosinophils infiltration changes between pre and post gluten free diet in Nonalcoholic Fatty Liver Disease Pediatric Celiac Disease Patients | Retrospective (years 2000-2023); 1 year of diet
  Duodenal eosinophils infiltration will be assessed in all historical subjects who had or did not have a change in liver steatosis degree between pre and post 1 year of gluten free diet, and who underwent gastroscopy both before and after start of gluten-free diet. Difference will be considered significant for p<0.05.
Body Mass Index changes between pre and post gluten free diet in Nonalcoholic Fatty Liver Disease Pediatric Celiac Disease Patients. | Retrospective (years 2000-2023); 1 year of diet
  Body mass index will be assessed in all historical subjects who had or did not have a change in liver steatosis degree between pre and post 1 year of gluten free diet. Difference will be considered significant for p<0.05.
Intestinal permeability markers changes in newly diagnosed Pediatric Celiac Disease Patients before and after gluten free diet: zonulin | 6 months [from T0 (before start of gluten-free diet) to T1 (after 6 months of gluten-free diet)]
  Zonulin serum levels changes will be assessed before and after 6 months of gluten free diet in newly diagnosed pediatric celiac disease patients both with and without liver steatosis. Difference will be considered significant for p<0.05.
  The assay will be carried out using the enzyme-linked immunosorbent assay method, with commercially available kits, following the manufacturers' instructions.
Intestinal permeability markers changes in newly diagnosed Pediatric Celiac Disease Patients before and after gluten free diet: occludin | 6 months [from T0 (before start of gluten-free diet) to T1 (after 6 months of gluten-free diet)]
  Occludin serum levels changes will be assessed before and after 6 months of gluten free diet in newly diagnosed pediatric celiac disease patients both with and without liver steatosis. Difference will be considered significant for p<0.05.
  The assay will be carried out using the enzyme-linked immunosorbent assay method, with commercially available kits, following the manufacturers' instructions.
Intestinal permeability markers changes in newly diagnosed Pediatric Celiac Disease Patients before and after gluten free diet: anti-occludin antibodies | 6 months [from T0 (before start of gluten-free diet) to T1 (after 6 months of gluten-free diet)]
  Anti-occludin antibodies serum levels changes will be assessed before and after 6 months of gluten free diet in newly diagnosed pediatric celiac disease patients both with and without liver steatosis. Difference will be considered significant for p<0.05. The assay will be carried out using the enzyme-linked immunosorbent assay method, with commercially available kits, following the manufacturers' instructions.
Intestinal permeability markers changes in newly diagnosed Pediatric Celiac Disease Patients before and after gluten free diet: claudin 1 | 6 months [from T0 (before start of gluten-free diet) to T1 (after 6 months of gluten-free diet)]
  Claudin 1 serum levels changes will be assessed before and after 6 months of gluten free diet in newly diagnosed pediatric celiac disease patients both with and without liver steatosis. Difference will be considered significant for p<0.05.
  The assay will be carried out using the enzyme-linked immunosorbent assay method, with commercially available kits, following the manufacturers' instructions.
Intestinal permeability markers changes in newly diagnosed Pediatric Celiac Disease Patients before and after gluten free diet: anti-claudin 1 antibodies | 6 months [from T0 (before start of gluten-free diet) to T1 (after 6 months of gluten-free diet)]
  Anti-claudin 1 antibodies serum levels changes will be assessed before and after 6 months of gluten free diet in newly diagnosed pediatric celiac disease patients both with and without liver steatosis. Difference will be considered significant for p<0.05.
  The assay will be carried out using the enzyme-linked immunosorbent assay method, with commercially available kits, following the manufacturers' instructions.
Duodenal mucosa damage markers changes in newly diagnosed Pediatric Celiac Disease Patients before and after gluten free diet: Intestinal Fatty Acid Binding Protein 2 | 6 months [from T0 (before start of gluten-free diet) to T1 (after 6 months of gluten-free diet)]
  Intestinal Fatty Acid Binding Protein 2 serum levels changes will be assessed before and after 6 months of gluten free diet in newly diagnosed pediatric celiac disease patients both with and without liver steatosis. Difference will be considered significant for p<0.05.
  The assay will be carried out using the enzyme-linked immunosorbent assay method, with commercially available kits, following the manufacturers' instructions.
Duodenal mucosa damage markers changes in newly diagnosed Pediatric Celiac Disease Patients before and after gluten free diet: lipopolysaccharide | 6 months [from T0 (before start of gluten-free diet) to T1 (after 6 months of gluten-free diet)]
  Lipopolysaccharide serum levels changes will be assessed before and after 6 months of gluten free diet in newly diagnosed pediatric celiac disease patients both with and without liver steatosis. Difference will be considered significant for p<0.05.
  The assay will be carried out using the enzyme-linked immunosorbent assay method, with commercially available kits, following the manufacturers' instructions.
Duodenal mucosa damage markers changes in newly diagnosed Pediatric Celiac Disease Patients before and after gluten free diet: lipopolysaccharide binding protein | 6 months [from T0 (before start of gluten-free diet) to T1 (after 6 months of gluten-free diet)]
  Lipopolysaccharide binding protein serum levels changes will be assessed before and after 6 months of gluten free diet in newly diagnosed pediatric celiac disease patients both with and without liver steatosis. Difference will be considered significant for p<0.05.
  The assay will be carried out using the enzyme-linked immunosorbent assay method, with commercially available kits, following the manufacturers' instructions.
Inflammatory markers changes in newly diagnosed Pediatric Celiac Disease Patients before and after gluten free diet: tumor necrosis factor a | 6 months [from T0 (before start of gluten-free diet) to T1 (after 6 months of gluten-free diet)]
  Tumor necrosis factor a levels changes will be assessed before and after 6 months of gluten free diet in newly diagnosed pediatric celiac disease patients both with and without liver steatosis. Difference will be considered significant for p<0.05.
  The measurement of inflammation markers will be performed by intracellular staining with flow cytometric method on peripheral blood mononuclear cells (PBMC) extracted from patients' blood samples.
Inflammatory markers changes in newly diagnosed Pediatric Celiac Disease Patients before and after gluten free diet: interleukin 1b | 6 months [from T0 (before start of gluten-free diet) to T1 (after 6 months of gluten-free diet)]
  Interleukin 1b levels changes will be assessed before and after 6 months of gluten free diet in newly diagnosed pediatric celiac disease patients both with and without liver steatosis. Difference will be considered significant for p<0.05.
  The measurement of inflammation markers will be performed by intracellular staining with flow cytometric method on peripheral blood mononuclear cells (PBMC) extracted from patients' blood samples.
Inflammatory markers changes in newly diagnosed Pediatric Celiac Disease Patients before and after gluten free diet: interleukin 6 | 6 months [from T0 (before start of gluten-free diet) to T1 (after 6 months of gluten-free diet)]
  Interleukin 6 levels changes will be assessed before and after 6 months of gluten free diet in newly diagnosed pediatric celiac disease patients both with and without liver steatosis. Difference will be considered significant for p<0.05.
  The measurement of inflammation markers will be performed by intracellular staining with flow cytometric method on peripheral blood mononuclear cells (PBMC) extracted from patients' blood samples.
Inflammatory markers changes in newly diagnosed Pediatric Celiac Disease Patients before and after gluten free diet: interleukin 12 | 6 months [from T0 (before start of gluten-free diet) to T1 (after 6 months of gluten-free diet)]
  Interleukin 12 levels changes will be assessed before and after 6 months of gluten free diet in newly diagnosed pediatric celiac disease patients both with and without liver steatosis. Difference will be considered significant for p<0.05.
  The measurement of inflammation markers will be performed by intracellular staining with flow cytometric method on peripheral blood mononuclear cells (PBMC) extracted from patients' blood samples.
Inflammatory markers changes in newly diagnosed Pediatric Celiac Disease Patients before and after gluten free diet: interleukin 18 | 6 months [from T0 (before start of gluten-free diet) to T1 (after 6 months of gluten-free diet)]
  Interleukin 18 levels changes will be assessed before and after 6 months of gluten free diet in newly diagnosed pediatric celiac disease patients both with and without liver steatosis. Difference will be considered significant for p<0.05.
  The measurement of inflammation markers will be performed by intracellular staining with flow cytometric method on peripheral blood mononuclear cells (PBMC) extracted from patients' blood samples.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Gastroenterological Paediatrics, Children's Hospital "G. Di Cristina", Palermo, Palermo
  - General Pediatrics Unit, Children's Hospital "G. Di Cristina", Palermo, Palermo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Husby S, Koletzko S, Korponay-Szabo IR, Mearin ML, Phillips A, Shamir R, Troncone R, Giersiepen K, Branski D, Catassi C, Lelgeman M, Maki M, Ribes-Koninckx C, Ventura A, Zimmer KP; ESPGHAN Working Group on Coeliac Disease Diagnosis; ESPGHAN Gastroenterology Committee; European Society for Pediatric Gastroenterology, Hepatology, and Nutrition. European Society for Pediatric Gastroenterology, Hepatology, and Nutrition guidelines for the diagnosis of coeliac disease. J Pediatr Gastroenterol Nutr. 2012 Jan;54(1):136-60. doi: 10.1097/MPG.0b013e31821a23d0. PMID 22197856
- [Background] Mansueto P, Spagnuolo G, Calderone S, D'Agate CC, Cosenza S, Leonardi G, Camilleri S, Pistone M, Seminara G, Alaimo C, Soresi M, Carroccio A, Garufi S. Improving the diagnostic approach to celiac disease: Experience from a regional network. Dig Liver Dis. 2022 Jun;54(6):771-775. doi: 10.1016/j.dld.2021.11.016. Epub 2021 Dec 21. PMID 34952810
- [Background] Al-Toma A, Volta U, Auricchio R, Castillejo G, Sanders DS, Cellier C, Mulder CJ, Lundin KEA. European Society for the Study of Coeliac Disease (ESsCD) guideline for coeliac disease and other gluten-related disorders. United European Gastroenterol J. 2019 Jun;7(5):583-613. doi: 10.1177/2050640619844125. Epub 2019 Apr 13. PMID 31210940
- [Background] Yoosuf S, Singh P, Khaitan A, Strand TA, Ahuja V, Makharia GK. Prevalence of Celiac Disease in Patients With Liver Diseases: A Systematic Review and Meta-Analyses. Am J Gastroenterol. 2023 May 1;118(5):820-832. doi: 10.14309/ajg.0000000000002123. Epub 2022 Dec 23. PMID 36599134
- [Background] Rinella ME, Lazarus JV, Ratziu V, Francque SM, Sanyal AJ, Kanwal F, Romero D, Abdelmalek MF, Anstee QM, Arab JP, Arrese M, Bataller R, Beuers U, Boursier J, Bugianesi E, Byrne CD, Castro Narro GE, Chowdhury A, Cortez-Pinto H, Cryer DR, Cusi K, El-Kassas M, Klein S, Eskridge W, Fan J, Gawrieh S, Guy CD, Harrison SA, Kim SU, Koot BG, Korenjak M, Kowdley KV, Lacaille F, Loomba R, Mitchell-Thain R, Morgan TR, Powell EE, Roden M, Romero-Gomez M, Silva M, Singh SP, Sookoian SC, Spearman CW, Tiniakos D, Valenti L, Vos MB, Wong VW, Xanthakos S, Yilmaz Y, Younossi Z, Hobbs A, Villota-Rivas M, Newsome PN; NAFLD Nomenclature consensus group. A multisociety Delphi consensus statement on new fatty liver disease nomenclature. Hepatology. 2023 Dec 1;78(6):1966-1986. doi: 10.1097/HEP.0000000000000520. Epub 2023 Jun 24. PMID 37363821
- [Background] Yodoshi T, Orkin S, Arce-Clachar AC, Bramlage K, Xanthakos SA, Valentino PL, Mouzaki M. Alternative Etiologies of Liver Disease in Children With Suspected NAFLD. Pediatrics. 2021 Apr;147(4):e2020009829. doi: 10.1542/peds.2020-009829. PMID 33785637
- [Background] Reilly NR, Lebwohl B, Hultcrantz R, Green PH, Ludvigsson JF. Increased risk of non-alcoholic fatty liver disease after diagnosis of celiac disease. J Hepatol. 2015 Jun;62(6):1405-11. doi: 10.1016/j.jhep.2015.01.013. Epub 2015 Jan 21. PMID 25617505
- [Background] Spadoni I, Zagato E, Bertocchi A, Paolinelli R, Hot E, Di Sabatino A, Caprioli F, Bottiglieri L, Oldani A, Viale G, Penna G, Dejana E, Rescigno M. A gut-vascular barrier controls the systemic dissemination of bacteria. Science. 2015 Nov 13;350(6262):830-4. doi: 10.1126/science.aad0135. PMID 26564856
- [Background] Wang HH, Lee DK, Liu M, Portincasa P, Wang DQ. Novel Insights into the Pathogenesis and Management of the Metabolic Syndrome. Pediatr Gastroenterol Hepatol Nutr. 2020 May;23(3):189-230. doi: 10.5223/pghn.2020.23.3.189. Epub 2020 May 8. PMID 32483543
- [Background] Hrncir T, Hrncirova L, Kverka M, Hromadka R, Machova V, Trckova E, Kostovcikova K, Kralickova P, Krejsek J, Tlaskalova-Hogenova H. Gut Microbiota and NAFLD: Pathogenetic Mechanisms, Microbiota Signatures, and Therapeutic Interventions. Microorganisms. 2021 Apr 29;9(5):957. doi: 10.3390/microorganisms9050957. PMID 33946843